CLINICAL TRIAL: NCT05692687
Title: A Prospective, Non-comparative, Multi-centre, Post-market Clinical Study to Evaluate the Safety and Performance of the Carbon Fibre Reinforced Polyetheretherketone Metatarso-Phalangeal (MTP) Plate (CoLink® PCR MTP Plate) for the Treatment of Hallux Rigidus
Brief Title: A Post-market Clinical Study to Evaluate the Safety and Performance of the Carbon Fibre Reinforced Polyetheretherketone Metatarso-Phalangeal (MTP) Plate (CoLink® PCR MTP Plate) for the Treatment of Hallux Rigidus
Status: Completed | Type: Observational
Sponsor: Invibio Ltd (Industry)
Collaborators: In2Bones (Unknown)
Responsible Party: Sponsor
Other Study IDs: IN2B01
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hallux Rigidus
MeSH Terms: conditions — Hallux Rigidus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical study involves the routine treatment of skeletally mature patients who have been diagnosed with hallux rigidus (stiffness of the first metatarso-phalangeal joint in the foot due to arthritis and degeneration of cartilage).

It follows standard practice surgery to treat this condition. This type of degenerative arthritis affects the joint of the big toe (hallux) which is attached to the foot. Taking part in this research will involve collecting data of the surgery to remove damaged cartilage and fix the two bones together with screws and a plate (called the CoLink® PCR MTP Plate).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years of age or older (> 18 years) and are skeletally mature.
2. Subjects who require surgical treatment for hallux rigidus and have been evaluated as appropriate candidates for treatment with the CoLink® PCR MTP Plate by the Investigator.
3. Subjects who, in the opinion of the Investigator, are able to understand this clinical study, co-operate with the procedures and are willing to return to the hospital for all the required post-operative follow-ups.
4. Subjects who are able to give voluntary, written informed consent to participate in this clinical study and from whom consent has been obtained.

Exclusion Criteria:

1. Subjects who have previously undergone MTP fusion surgery or implant arthroplasty in the foot to be treated.
2. Subjects who require bi-lateral MTP fusion surgery.
3. Subjects with evidence of tumour and/or malignant disease with resultant life expectancy of less than two years.
4. Subjects with a known allergy to the material used in the instrumentation.
5. Subjects with evidence of an active infection and/or with any condition that would compromise their participation and follow-up in this clinical study.
6. Subjects who have any conditions outlined as contraindicated in the Instructions for Use.
7. Female subjects who are pregnant or lactating.
8. Subjects who are known drug or alcohol abusers, or with a baseline opioid use greater than 30 mg of morphine equivalent/day, or with psychological disorders that could affect follow-up care or treatment outcomes.
9. Subjects who are current smokers or have stopped smoking less than 6 months ago.
10. Subjects who are currently enrolled in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective study so patients taken from those undergoing treatment surgery for Hallux Rigidus.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Bone Fusion | 6 months
  Successful radiographic union: where union is defined as 'evidence of bridging' between the metatarsal bone and proximal phalanx bone by an independent imaging company.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - South Florida Foot and Ankle Center, Lake Worth, Florida
  - University of Kansas Medical Centre, Kansas City, Kansas
  - Mississippi Sports Medicine and Orthopedic Center,, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No